CLINICAL TRIAL: NCT05310396
Title: Efficacy of a Nutrient Blend Comprised of Specific Nutrients in Improving Neurocognitive and Behavioural Outcomes in Infants: a Randomized, Controlled, Intervention Study
Brief Title: Efficacy of a Nutrient Blend in Improving Neurocognitive and Behavioral Outcomes in Infants: a Randomized, Controlled, Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20.26.INF
Record Dates: First submitted 2022-01-04; First posted 2022-04-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Infant Nutrition; Cognitive Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powdered cow's milk-based infant formula containing uniquely processed whey protein (Experimental): Starter and follow up formula containing combination of an HMO blend, myelin nutrient blend, and MOS
  Interventions: Other: Experimental formula
- Powdered infant fortified cow's milk (Active Comparator): Standard Starter and follow up formula without added HMOs or MOS containing lower levels of myelin nutrients
  Interventions: Other: Control Formula

INTERVENTIONS:
Other: Experimental formula — Cow's milk-based infant formula with a specific blend of nutrients at pre-defined levels
  Arms: Powdered cow's milk-based infant formula containing uniquely processed whey protein
Other: Control Formula — Cow's milk-based infant formula with standard nutritional composition
  Arms: Powdered infant fortified cow's milk

SUMMARY:
The purpose of this study is to demonstrate the efficacy of the nutrient blend in a starter infant formula (IF) and follow up infant formula (FUF) in improving the neurocognitive and behavioural outcomes among formula-fed infants randomized to the experimental formula (EF) versus the control formula (CF).

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, double-blind, 2-arm parallel-group clinical trial in the Philippines. Subjects will be recruited from a single centre; in case of insufficient recruitment, more sites will be added to the study. The clinical trial is composed of two parts: a double-blind interventional period and a follow-up period. The first period is the double-blind intervention phase from enrolment (V1) until age 12 months (V5). The intervention will be provided only during this double-blind phase. The second period is a non-interventional follow-up period from age 12 months until age 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Infants between 45 to 60 days of age at enrolment
2. Infant's ≥ 37 completed weeks of gestation, with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg and singleton born.
3. Infants generally healthy at birth with an Apgar score ≥7 at 5 min
4. Exclusively formula fed for at least 14 days before randomization and the choice of formula feeding has been taken by the parents before the beginning of the trial
5. Signed informed consent obtained for infant's and parents' participation in the study
6. Parents of infant agree not to enrol infant in another interventional clinical research study while participating in this study
7. Parent of infant agrees to provide to their infants the study formula and not replace it with another commercial formula.
8. Parent of the infant is of legal age of consent, must understand the informed consent form and other study documents, willing and able to fulfil the requirements of the study protocol.
9. Parent of infant can be contacted directly by telephone or email throughout the study.

Exclusion Criteria:

1. History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant.
2. Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion)
3. Infants with known or suspected intolerance to cow milk infant formula or allergy
4. The infant is identified to have a chromosomal or major congenital anomaly or significant medical and/or genetic conditions that interferes with adequate functioning in daily life or likely to interfere with normal growth and development or with the normal maturation of visual or cognitive function (including visual/hearing impairment), known head or brain disease, injury such as microcephaly or macrocephaly, immunocompromised or suffered from significant illness, developmental delay or disability
5. Infants who have been adopted or are foster infants
6. Infants born to mothers with chronic illness, such as HIV disease, renal or hepatic disease, type 1 or type 2 diabetes, alcoholism, or substance abuse
7. Presence of a first degree relative with neurologic or psychiatric diseases (e.g., attention deficit hyperactivity disorder, autism, behavioural problems, bipolar disorder, depression, intellectual disability, or schizophrenia).

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Scores on the Cognitive subscale of the Bayley Scale of Infant Development, 4th Edition | 12 months
  Change in the scores on the Cognitive subscale. The scores range from 40 to 160 and higher scores indicate a better cognitive outcome

SECONDARY OUTCOMES:
Infant Global developmental status in all domains of the Bayley Scale of Infant Development, 4th Edition | 6 months, 9 months, 12 months, and 24 months
  Infant Language, motor, socio-emotional, adaptive behaviour, and cognitive scores will be assessed
Infant Visual attention | 4 months, 6 months, 9 months, and 12 months
  Developmental status of infants' visual attention will be assessed using the infant Gap-Overlap task
Infant Visual learning | 4 months, 6 months, 9 months, and 12 months
  Infant's quality of attention will be assessed using the infant visual habituation task as augmented with heart rate
Early language development | Words and Gestures (long form) at 12 months and Words and Sentences (long form) at 24 months
  Assessed using the MacArthur-Bates Communicative Development Inventories
Working memory and inhibitory control | 24 months
  Assessed using the A-not-B Invisible Displacement Task
Behavioral manifestations of executive function | 24 months
  Assessed using the Behavior Rating Inventory of Executive Function-Preschool version. The questionnaire consists of scales such as Inhibit, Shift, Emotional Control, working memory, plan and organize and Indexes such as Inhibitory Self control, Flexibility Index, Emergent metacognition index and Global Executive Composite. T scores are used to interpret the child's level of executive functioning on the BRIEF-P. scores provide information about a child's scores relative to the scores of children in the standardization sample
Infant temperament | 1.5-2 months, 6 months, and 12 months
  Assessed using the Infant Behaviour Questionnaire Revised Short Form. The questionnaire assess dimensions of temperament along 14 scales on a 7-point Likert scale on behavior occurrence, with 1 being never and 7 being always (Activity level, Distress to limitations, Approach, Fear, Duration of orienting, smiling and laughter, vocal reactivity, Sadness, Perceptual sensitivity, High-intensity pleasure, Low-intensity pleasure, Cuddliness, Soothability, Falling Reactivity/Rate of Recovery From Distress)
Child temperament | 24 months
  Child temperament will be assessed using the Early Childhood Behavior Questionnaire- Short Form. The questionnaire measures 18 discrete traits embedded within three higher-order factors on a 7-point Likert scale on behavior occurrence, with 1 being never and 7 being always. Negative Affect (Discomfort, Fear, Frustration, Motor Activation, Sadness, Perceptual Sensitivity, Shyness, Soothability), Surgency (Impulsivity, Activity Level, High Intensity Pleasure, Sociability, Positive Anticipation), and Effortful Control (Inhibitory Control, Attention Shifting, Low Intensity Pleasure, Cuddliness, and Attentional Focusing).
Infant sleep | 1.5-2 months, 6 months, 12 months, and 24 months
  Infant daytime and night-time sleep patterns, parent perception, and sleep-related behaviours will be assessed using the Brief Infant Sleep Questionnaire
Infant fecal microbiota | 1.5-2 months (but before starting study formula), and just prior to 6 months, and 12 months
  Overall fecal microbiota composition, diversity, microbiota community types will be assessed using next generation sequencing (NGS) technology
Infant immune and gut health biomarkers | 1.5-2 months (but before starting study formula), 6 months, and 12 months
  Fecal markers of immune and gut barrier, such as but no restricted to total secretory IgA (sIgA), lipocalin-2, calprotectin, and α-1-antitrypsin will be assessed by ELISA

OTHER OUTCOMES:
Infant GI Tolerance | 1.5-2 months, 6 months, and 12 months
  Assessed using Infant Gastrointestinal Symptom Questionnaire. The questionnaire comprises of 13 questions assessed on a 5-point Likert Scale with overall scores of 13 (best) to 65 (worst) for overall GI symptoms
Toddler GI Tolerance | 24 months
  Assessed using Toddler Gut Comfort Questionnaire. The questionnaire comprises of 10 questions assessed on a 6-point scale for frequency and severity, ranging from 1 (None or Not at all) to 6 (Always or Very strong).
Head circumference | 1.5-2 months, 4 months, 6 months, 9 months, 12 months and 24 months
  Head circumference measured in cm
Weight | 1.5-2 months, 4 months, 6 months, 9 months, 12 months and 24 months
  Weight measured in grams
Length/Height | 1.5-2 months, 4 months, 6 months, 9 months, 12 months and 24 months
  Length/Height measured in cm
BMI | 1.5-2 months, 4 months, 6 months, 9 months, 12 months and 24 months
  Weight and height will be combined to report BMI in kg/m2
Z-scores | 1.5-2 months, 4 months, 6 months, 9 months, 12 months and 24 months
  Weight-for-age, height-for-age, weight-for-height, head circumference-for-age, BMI-for-age, weight and height velocity
Incidence of infant illness and infection | 1.5-2 months, 13 months, and additionally at 23.8 months and 24 months
  Collected as part of standard adverse events reporting for safety assessment including medication use and paper Infant Illness Diary continuously from enrolment until V5 (12 mo).
Formula intake adherence | Completed by the parent on a weekly basis beginning on the first day of intervention (1 day after V1 after the stool collection)
  Assessed using Study Compliance Diary
Infant dietary intake | Completed at home just prior to clinic visits at 6 months, 12 months and 24 months
  Will be assessed using a 24-hour Dietary Recall completed by the parent / caregiver
Maternal Postpartum depression/ anxiety | 1.5-2 months and 4 months
  Assessed using an Edinburgh Postnatal Depression Scale. The questionnaire comprises of 10 questions. Responses are scored 0, 1, 2 and 3 based on the seriousness of the symptom. The total score is obtained by adding together the scores for each of the 10 items. Scores above 12 or 13 are likely to be indicative of possible depression
Parenting Stress | 1.5-2 months, 6 months, 12 months and 24 months
  Assessed using a Parenting Stress Index-Short Form. The questionnaire comprises of thirty-six items divided into three domains: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC), which combine to form a Total Stress scale. Each subscale consists of 12 items rated from 1 (strongly disagree) to 5 (strongly agree), with subscales scores ranging from 12 to 60. A Total score is calculated by summing the three subscales scores, ranging from 36 to 180. Scores of 90 or above may indicate a clinical level of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, MD, Principal Investigator — Las Pinas Doctors Hospital
Locations (1):
- Las Piñas Doctors Hospital, Las Piñas, Philippines

IPD SHARING:
Plan to Share IPD: No